CLINICAL TRIAL: NCT06409104
Title: Propofol Versus Dexmedetomidine for Sedation of Cancer Patients Undergoing Endoscopic Retrograde Cholangio-Pancreatography: Randomized Single Blinded Controlled Study
Brief Title: Propofol Versus Dexmedetomidine for Sedation of Cancer Patients Undergoing ERCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MS-211-2023
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Sedation in ERCP
Keywords: ERCP; Endoscopic; cancer; sedation; propofol; Dexmedetomidine
MeSH Terms: conditions — Neoplasms | interventions — Propofol; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: * To compare hemodynamic profile of dexmedetomidine and Propfol during sedation in patients undergoing ERCP.
  * To study both agents effect on respiratory complications.
  * To demonstrate the effect of both drugs on cognitive functions.
  * To assess the effect of both drugs on duration of procedure and number of interruptions.
Who Masked: Participant, Investigator
Masking Description: The patients will be randomly assigned into two equal comparable groups using computer- generated random numbers in opaque closed envelopes, each of which will include 101 patients. Randomization will be done by statistician and each group of the patient will revealed only when the included patient is transferred to preanesthetic room.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol (Active Comparator): will receive 1-2 mgkg-1 propofol injection over 30s followed by of propofol a 0.05 to 0.1 mg /kg/min infusion .
  Interventions: Drug: Propofol
- Dexmedetomidine (Active Comparator): will receive dexmedetomidine at a loading dose of 1 μg/kg over 10 min, followed by a 0.2-0.7-μg/kg/h infusion.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Propofol — will receive 1-2 mgkg-1 propofol injection over 30s followed by of propofol a 0.05 to 0.1 mg /kg/min infusion
  Arms: Propofol
Drug: Dexmedetomidine — will receive dexmedetomidine at a loading dose of 1 μg/kg over 10 min, followed by a 0.2-0.7-μg/kg/h infusion.
  Arms: Dexmedetomidine

SUMMARY:
The aim of this study is to compare the efficacy and safety of propofol and dexmedetomidine during ERCP regarding hemodynamic, respiratory, sedative and cognitive functions.

DETAILED DESCRIPTION:
Endoscopic retrograde cholangiopancreatography (ERCP) plays a crucial role in the diagnosis and treatment of pancreaticobiliary pathologies, and its use has increased in recent years. The procedure lasts from 30 to 60 position. Patients usually cannot tolerate the procedure because of pain, uncomfortable position, fear, and nausea without adequate sedation; therefore, ERCP is generally performed under moderate to deep sedation or even GA. ERCP under general anesthesia has several limitations. The procedure is often prolonged due to extra time required for patient preparation, induction of anesthesia, tracheal intubation, and recovery. In addition, the cost per procedure is higher. Deep sedation, on the other hand, is an alternative that is used by specific centers under anesthesiologist supervision instead of general anesthesia. Deep sedation has the advantage of offering the extra time required for general anesthesia and better procedure conditions in relation to conscious sedation.

Propofol is a popular drug that is frequently used in day surgery because of its early onset activity, short duration of action, and the fact that the patient regains normal mental functions only minutes after intravenous application. However, an increased dose of propofol may cause undesirable side effects such as hypoxia which is a common occurrence during upper GI endoscopy under sedation with propofol prolonged hypoxia is the most common cause of cardiac arrhythmia and coronary ischemia .Also, propofol lacks adequate analgesic effects to inhibit visceral traction, pain other side effects of propofol include hypotension and apnea.

In recent years, dexmedetomidine has been used as an alternative to Propofol in conscious sedation applications. Because it provides sedation and analgesia but does not cause respiratory depression, dexmedetomidine is considered a suitable drug for operations that are performed under local anesthesia.

According to authors best knowledge, there are no enough studies comparing both drugs in patients undergoing ERCP

Aim of the work The aim of this study is to compare the efficacy and safety of propofol and dexmedetomidine during ERCP regarding hemodynamic, respiratory, sedative and cognitive functions.

Objectives:

* To compare the hemodynamic profile of dexmedetomidine and Propofol during sedation in patients undergoing ERCP.
* To study both agents effect on respiratory complications.
* To demonstrate the effect of both drugs on cognitive functions.
* To assess the effect of both drugs on the duration of the procedure and the number of interruptions.

Hypothesis:

The investigators hypothesize that dexmedetomidine will provide better sedation and analgesia with fewer side effects when compared to propofol in patients undergoing ERCP.

ELIGIBILITY:
Inclusion Criteria:

* Age starting from 21 to 60 years.
* Genders eligible for study: males and females
* ASA II-III
* Undergoing ERCP
* 18.5 to 30 kg/m2

Exclusion Criteria:

* Patient refusal
* Known allergy to drugs used in the study.
* Use of any anti-coagulants
* Neurological disorders
* Advanced liver or kidney disease
* Patient with psychiatric disorders

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 202 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Bispectral Index sedation Score | intraoperative
  >90 indicates an awake patient; 71-90, mild to moderate sedation; 61-70, deep sedation; and 40-60, general anesthesia

SECONDARY OUTCOMES:
Change in heart rate during procedure | intraoperative
  Change in heart rate during procedure
Change in MAP | intraoperative
  Change in MAP during procedure
Pain during procedure according to Facial Pain Rating Scale | first 2hours postoperative
  Pain during procedure according to Facial Pain Rating Scale (FPS;0 no pain-10 maximum pain)
Duration to recovery after the end of procedure | first 2hours postoperative
  Duration to recovery after the end of procedure
Total doses of both agents used | intraoperative
  Total doses of Propofol or Dexmedetomidine used

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Mohamed Soliman, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
after publication